CLINICAL TRIAL: NCT05013385
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Phase IIa Trial to Evaluate Spesolimab (BI 655130) Efficacy in Patients With Fibrostenotic Crohn's Disease
Brief Title: A Study to Test Whether Spesolimab Helps People With Crohn's Disease Who Have Symptoms of Bowel Obstruction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1368-0059; 2020-005770-99 (EudraCT Number)
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Fibrostenotic Crohn´s Disease
MeSH Terms: interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spesolimab (Experimental)
  Interventions: Drug: Spesolimab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spesolimab — Spesolimab
  Arms: Spesolimab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to adults, between 18 and 75 years of age, who have narrowings in the small bowel (strictures) due to Crohn's disease. Strictures can lead to bowel obstruction (blockage). People whose symptoms got worse because of strictures can join the study. Participants get standard treatment for Crohn's disease and the strictures. The purpose of the study is to test whether the strictures improve further when treated with a medicine called spesolimab added to standard treatment.

Participants are in the study for about 1 year and 4 months. In the first 3 months, participants get standard treatment only. After 3 months, participants whose condition improved are put into 2 groups randomly, which means by chance. One group gets spesolimab added to their standard treatment. The other group gets placebo added to their standard treatment. Both spesolimab and placebo are given as infusions into a vein. Placebo infusions look like spesolimab infusions but do not contain any medicine. For the first 2 months, participants get the infusions every month. Thereafter, participants get the infusions every 2 months.

During the study, participants have about 11 visits to the study site. The doctors regularly check participants' health and take note of any unwanted effects. At 3 of the visits, doctors take images of the bowel using Magnetic Resonance Imaging and with an endoscope. At these visits, the doctors also take a small sample of bowel tissue (biopsy). The participants note their symptoms of Crohn's disease and how the symptoms affect daily life in an electronic diary. At the end of the study, results from the diaries and bowel imaging are compared between the spesolimab group and the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of legal age
* Established diagnosis of clinical Crohn's Disease
* Suspicion of symptomatic small bowel obstruction at screening
* 1 or 2 naïve or anastomotic stenoses in the terminal ileum, with at least one being in reach of ileocolonoscopy as defined by the CrOhN´S disease antifibrotic STRICTure Therapies (CONSTRICT) criteria, confirmed by MRE
* Have achieved a Symptomatic Stenosis Response after optimized anti-inflammatory therapy
* Absent, mild or moderate endoscopic activity defined by Simple Endoscopic Score in Crohn's Disease (SES-CD) ≤12 Further criteria apply

Exclusion Criteria:

* More than 2 small intestinal stenoses
* No stenosis is in reach of ileocolonoscopy
* Patients who require immediate endoscopic balloon dilation or surgical intervention as per the investigator´s discretion or who have undergone any of the two within the 6 months prior to the study
* Failure of >2 different biological drug classes
* Current complications of Crohn's Disease such as enterocutaneous, internal or rectovaginal fistules, short gut syndrome or abscess,
* Use of any prohibited concomitant medications as described in the study protocol
* Active tuberculosis (TB) or history of latent TB that has not been treated Further criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Washington University School of Medicine, St Louis, Missouri, United States
- Heritage Medical Research Clinic, Calgary, Alberta, Canada
- Kitasato Institute Hospital, Tokyo, Minato-ku, Japan
- Sahlgrenska Universitetssjukhuset, Mölndal, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was designed to have a Lead-in Period where background medication is optimized, a Randomized Blinded Treatment Period and a Follow-up Period. At the end of the Lead-in Period, if eligibility criteria were fulfilled patients would have been randomized to either spesolimab (BI 655130) or placebo for the blinded treatment period.
  The trial was terminated when only 5 patients had entered the lead-in period. No patient was randomized and received spesolimab or placebo.
Pre-assignment Details: All subjects who entered the Lead-in period were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Enrolled Patients: Fibrostenotic Crohn's Disease patients who were eligible to enter the Lead-In period of the trial were planned to receive during the Lead-In Period standard medical treatment which included 2 weeks of corticosteroids to be tapered according to a standardized 8 week regimen and individual optimization of anti-inflammatory biological treatment. After 8 weeks of optimized biological anti-inflammatory therapy would have been completed, only patients who would have achieved a Symptomatic Stenosis Response and an absent or mild-to-moderate colonic endoscopic activity (colonic Simple Endoscopic Score in Crohn's Disease (SES-CD) ≤12) would have been eligible for randomization into the Blinded Treatment Period.
Period: Overall Study
Arm/Group | Enrolled Patients
Started (Patients who entered the Lead-In Period) | 5
Patients Who Entered the Randomized Blinded Treatment Period | 0
Completed | 0
Not Completed | 5
Not completed — Sponsor's decision to terminate the trial | 5

BASELINE CHARACTERISTICS:
Population: Enrolled patients: Fibrostenotic Crohn's Disease patients who were eligible to enter the Lead-In period of the trial.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Maintained Symptomatic Stenosis Response at Week 48
Time Frame: At Week 48.
Population: Study was terminated early. 5 patients entered the Lead-In Period but no patient entered the Randomized Blinded Treatment Period and received the investigational medical products (spesolimab or placebo). Outcome Measures were planned to be reported for the Randomized Blinded Treatment Period.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 0

2. Primary Outcome: Proportion of Patients With Radiographic Stenosis Response at Week 48
Time Frame: At Week 48.
Population: as for outcome 1
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Patients With Maintained Symptomatic Stenosis Response at Week 24
Time Frame: At Week 24.
Population: as for outcome 1
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Patients With Radiographic Stenosis Response at Week 24
Time Frame: At Week 24
Population: as for outcome 1
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events data were planned to be reported for the Randomized Blinded Treatment Period. Since no patient was randomised to receive the investigational medical products (spesolimab or placebo) the number of participants at risk for "All-Cause Mortality", "Serious Adverse Events" and "Other Adverse Events" equals "0". The "0" in the All-Cause Mortality, Serious Adverse Events, and "Other Adverse Events" sections refers to "Not applicable".
Arm/Group | Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT05013385/Prot_SAP_000.pdf